CLINICAL TRIAL: NCT07250750
Title: A Phase 1b/2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Investigate A) the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of IM-101 in Adult Participants With Generalized Myasthenia Gravis, and B) the Efficacy and Safety of Treatment of IM-101 in Adult Participants With Generalized Myasthenia Gravis and Ocular Myasthenia Gravis
Brief Title: A Phase 1b/2 Study of IM-101 in Adult Participants With Generalized Myasthenia Gravis and Ocular Myasthenia Gravis
Acronym: Synergy-MG
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmunAbs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM-101_MG_2.1; 2025-522406-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-26; First posted 2025-11-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Myasthenia Gravis
Keywords: IM-101; Myasthenia Gravis; C5 inhibitor
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A MAD Cohort 1 (Experimental): IM-101 Low dose or Placebo
  Interventions: Drug: IM-101 Part A; Drug: Placebo Part A
- Part A MAD Cohort 2 (Experimental): IM-101 Mid dose or Placebo
  Interventions: Drug: IM-101 Part A; Drug: Placebo Part A
- Part A MAD Cohort 3 (Experimental): IM-101 High dose or Placebo
  Interventions: Drug: IM-101 Part A; Drug: Placebo Part A
- Part A MAD Cohort 4 (Optional) (Experimental): IM-101 or Placebo if additional dose is needed per IDMC decision
  Interventions: Drug: IM-101 Part A; Drug: Placebo Part A
- Part B Expansion AChR positive gMG (Experimental): IM-101 or Placebo
  Interventions: Drug: IM-101 Part B; Drug: Placebo Part B
- Part B Expansion AChR negative gMG (Experimental): IM-101 or Placebo
  Interventions: Drug: IM-101 Part B; Drug: Placebo Part B
- Part B Expansion oMG (Experimental): IM-101 or Placebo
  Interventions: Drug: IM-101 Part B; Drug: Placebo Part B

INTERVENTIONS:
Drug: IM-101 Part A — Participants will receive IM-101 intravenously (IV), at a loading dose on Day 1 and Day 15 followed by maintenance dose and Day 29.
  Arms: Part A MAD Cohort 1; Part A MAD Cohort 2; Part A MAD Cohort 3; Part A MAD Cohort 4 (Optional)
Drug: Placebo Part A — Participants will receive Placebo intravenously (IV), at a loading dose on Day 1 and Day 15 followed by maintenance dose on Day 29.
  Arms: Part A MAD Cohort 1; Part A MAD Cohort 2; Part A MAD Cohort 3; Part A MAD Cohort 4 (Optional)
Drug: IM-101 Part B — Participants will receive IM-101 intravenously (IV), at a loading dose on Day 1 and Day 15 followed by maintenance dose on Day 29, D57 and D85.
  Arms: Part B Expansion AChR negative gMG; Part B Expansion AChR positive gMG; Part B Expansion oMG
Drug: Placebo Part B — Participants will receive Placebo intravenously (IV), at a loading dose on Day 1 and Day 15 followed by maintenance dose on Day 29, D57 and D85.
  Arms: Part B Expansion AChR negative gMG; Part B Expansion AChR positive gMG; Part B Expansion oMG

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and potential efficacy of IM-101 in adult participants with AChR antibody-positive gMG. Subsequently, the safety and efficacy of the selected IM-101 dose-regimen will be tested in participants with AChR antibody-negative gMG and participants with AChR antibody-positive or AChR antibody-negative oMG.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide signed informed consent
2. Willingness to consent to screening for genetic muscular diseases
3. Male or female aged ≥ 18 years and < 75 years
4. Diagnosed with MG
5. On a stable dose of background therapy for the treatment of MG
6. Body weight ≥ 40 kg at screening
7. Vaccinated against meningococcal infection (Neisseria meningitidis), streptococcus pneumoniae, and haemophilus influenzae type B

Exclusion Criteria:

1. Previous exposure to IM-101
2. Anti-MuSK antibody Positive
3. History of malignant thymoma, or history of cancer within the past 5 years of screening
4. History of N. meningitidis infection
5. Has been treated with any complement inhibitor, but failed due to intolerability or lack of efficacy

Full eligibility criteria is available in the study protocol.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
[Part A] Incidence of TEAEs, SAEs, AEs that led to premature discontinuation, and AESIs across 3 ascending dose regimens (each with 3 administrations) in participants with AChR antibody-positive gMG | From first dose of study drug (Day 1) up to 70 days after the last dose of study drug, up to approximately 99 days.
  An AE is any untoward medical occurrence in a clinical study participant administered with a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important. Treatment-emergent AEs associated with a. Grade > 2 hypersensitivity or IRR, b. Infection c. Any potential kidney failure and d. Any potential Hy's Law case (> 3 × ULN of either ALT/AST with concurrent > 2 × ULN of total bilirubin and lack of alternate etiology) will be considered AESIs.
[Part B] Incidence of TEAEs, SAEs, AEs that led to premature discontinuation, and AESIs of IM-101, compared with placebo, in participants with AChR antibody-positive gMG, AChR antibody-negative gMG, and oMG | From first dose of study drug (Day 1) up to 84 days after the last dose of study drug, up to approximately 169 days.
  An AE is any untoward medical occurrence in a clinical study participant administered with a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important. Treatment-emergent AEs associated with a. Grade > 2 hypersensitivity or IRR, b. Infection c. Any potential kidney failure and d. Any potential Hy's Law case (> 3 × ULN of either ALT/AST with concurrent > 2 × ULN of total bilirubin and lack of alternate etiology) will be considered AESIs.
[Part B] Change from baseline to Week 16 in the Myasthenia Gravis-Activities of Daily Living (MG-ADL) Total Score for gMG cohorts | Baseline, Week 16
  Change from baseline in MG-ADL total score over 16 Weeks will be reported. The MG-ADL provides a rapid assessment of the participant's MG symptom severity. Eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, eyelid droop) are rated on a 4-point scale: 0 (no impairment) to 3 (severe impairment). The total score will be sum of eight function scores and can range from 0 to 24. A higher score indicates greater symptom severity.
[Part B]Change from baseline to Week 16 in Myasthenia Gravis Impairment Index (MGII) ocular score for oMG cohorts | Baseline, Week 16
  Change from baseline in MGII ocular score over 16 Weeks will be reported. The MGII is a scoring tool measuring disease severity. It consists of 22 patient-reported outcomes (PRO) and 6 physical examinations (PE). The Ocular PRO score varies between 0 and 18. The higher the score, the more severe the disease.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (8):
  - Neurology of Central Florida Research Center, LLC, Altamonte Springs, Florida
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Missouri
  - Nerve & Muscle Center of Texas, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
- Bulgaria (5):
  - Medical Center Hera - branch Montana, Montana
  - "MHAT Avis - Medica" OOD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - Haelan Care 4 Medical Center EOOD, Varna
- Italy (3):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia, Brescia
  - Ospedale San Raffaele, Milan, Milano
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Milano
- Poland (5):
  - Neurologia Slaska Centrum Medyczne, Katowice
  - Twoja Przychodnia NCM, Nowa Sól
  - Twoja Przychodnia PCM, Poznan
  - NZOZ Neuro-Kard Ilkowski i Partnerzy Spółka Partnerska Lekarzy, Poznan
  - Samodzielny Publiczny Szpital Kliniczny nr 1 im. Prof. Stanislawa Szyszko, SUM, Zabrze
- General Hospital MSB Medical System Belgrade, Belgrade, Serbia
- Spain (3):
  - Hospital Universitario Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre